CLINICAL TRIAL: NCT03816384
Title: Effect of Active Drain Line Clearance With or Without Silver on Catheter-Associated Bacteriuria (The CAB Study)
Brief Title: Effect of Active Drain Line Clearance on Catheter-Associated Bacteriuria
Acronym: CAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Declined to pursue Study due to anticipated low enrollment numbers
Sponsor: Potrero Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRD-06-100548
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Critical Illness; Burns; Surgery; Urinary Tract Infections; Bacteriuria
Keywords: urinary catheter
MeSH Terms: conditions — Critical Illness; Burns; Urinary Tract Infections; Bacteriuria

STUDY DESIGN:
Intervention Model Description: Multi-center, Randomized-Controlled-Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Standard of Care (Active Comparator): Patients will receive Standard of Care, commercially available catheter utilized by hospital system.
  Interventions: Device: Standard of Care
- Drain Line Clearance (DLC) Group (Experimental): Patients will receive FDA-approved Accuryn Monitoring System with active drain line clearance and plain silicone catheter.
  Interventions: Device: DLC Group
- Drain Line Clearance and Silver (DLCS) Group (Experimental): Patients will receive FDA-approved Accuryn Monitoring System with active drain line clearance and silver-doped silicone catheter.
  Interventions: Device: DLCS Group

INTERVENTIONS:
Device: Standard of Care — Standard of care urinary drainage system.
  Arms: Standard of Care
Device: DLC Group — Urinary drainage system with active drain line clearance and plain silicone catheter.
  Arms: Drain Line Clearance (DLC) Group
Device: DLCS Group — Urinary drainage system with active drain line clearance and silver-doped silicone catheter.
  Arms: Drain Line Clearance and Silver (DLCS) Group

SUMMARY:
Catheter-associated urinary tract infections (CAUTI) are the most common nosocomial infections in critically ill patients and are responsible for high morbidity rates, increased hospital stays and associated costs.

The purpose of this study is to evaluate whether active drain line clearance by the Accuryn Monitoring System reduces the incidence of CAUTI in hospitalized patients requiring catheters.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is the most common healthcare associated infection (HAI) acquired in hospitals and is estimated to account for approximately 13% of hospital infections in the United States, of which 75% are associated with indwelling urinary catheters. It is estimated that between 12-16% adult inpatients will receive an indwelling urinary catheter during their hospital stay. The rate of catheter-associated UTI (CAUTI) are highest in burn ICUs, followed by inpatient medical wards and neurosurgical ICUs.

The purpose of this study is to evaluate whether active drain line clearance by the Accuryn Monitoring System reduces the incidence of bacteriuria and/or CAUTI in patients requiring catheters for more than 72 hours. This study will also evaluate the efficacy in reducing bacteriuria of the Accuryn silver fabricated silicone catheters.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥ 18)
2. Patient or Legally Authorized Representative (LAR) possess the capacity to provide informed consent
3. Indication for a urinary bladder catheter (or one currently in place)
4. Expected urinary catheter requirement ≥ 72 hours
5. No current urinary tract infection
6. No current indication for prophylactic antibiotics. If a surgical patient, receive perioperative antibiotics for no greater than 24 hours

Exclusion Criteria:

1. Inability to receive a urinary bladder catheter
2. Chronic suprapubic catheter in place
3. Expected survival < 72 hours
4. Receipt of systemic antibiotics within 48 hours of enrollment, other than prophylactic antibiotics given at the time of surgery
5. Surgery of the genitourinary tract in the past 6 months prior to admission
6. Deemed unfit for the protocol by the investigator for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in percentage of catheter-associated bacteriuria | 30 days
  To study the difference in rate of catheter-associated bacteriuria between SOC catheters and Accuryn silicone or Accuryn silver-doped catheters with active drain line clearance.

SECONDARY OUTCOMES:
Percentage of asymptomatic (ASB) and symptomatic (CAUTI) bacteriuria | 30 days
  To study the incidence and progression of asymptomatic bacteriuria and CAUTI in patients with prolonged foley catheters for greater than 72 hours.
Time to Bacteriuria (ASB and CAUTI) | 30 days
  To study the progression of asymptomatic bacteriuria and CAUTI in patients with prolonged foley catheters for greater than 72 hours.
Urine Culture Comparisons | 30 days
  To study the correlation between patient urine cultures and cultures taken from the Foley (Foley tip, urine sampled from collection bag).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Foster, MD, Principal Investigator — Maricopa Integrated Health System (MIHS)

IPD SHARING:
Plan to Share IPD: No